CLINICAL TRIAL: NCT06824584
Title: Relationship Between Physical Fitness and Psychopathology, Cognition and Quality of Life in Patients Diagnosed With Schizophrenia: a Mixed Method Study.
Acronym: COFESQ
Status: Active, not recruiting | Type: Observational
Sponsor: Universidade da Coruña (Other)
Collaborators: Servicio Gallego de Salud (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024/013
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia and Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; physical fitness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the physical fitness and the influence of possible factors (disease symptomatology, cognitive status, patient functioning and degree of perceived quality of life) on patients diagnosed with schizophrenia and schizoaffective disorder older than 18 years in an outpatient setting. The main question it aims to answer is:

Do the symptoms of the illness influence the level of physical fitness of patients?

Participants will complete a series of questionnaires assessing their cognitive status, perceived quality of life and disease severity, and physical activity assessments to measure their cardiovascular endurance and muscular power.

DETAILED DESCRIPTION:
A mixed-methods research design will be carried out. Two different study designs will be used:

- Stage 1: Cross-sectional study: During the first 3 months, recruitment will start. This task will be carried out by the nurses of the mental health unit and by the director of the psycho-social and labor rehabilitation center of the Alume association, located in Lugo. If the patient agrees to participate, he or she will have to give written consent by signing the patient information sheet provided. If the patient has a legal representative, he or she should also provide written informed consent. Over the next 3 months, participants will be evaluated. Principal investigator will contact them via telephone or online texting (depending on each participant's individual choice) to meet them at the gym where the research team will conduct patients' assessments. An initial anamnesis will be performed containing questions related to the patient's sociodemographic data and to questions related to their illness. Along with this first step, anthropometric measurements will be taken for each individual, both with manual measurements. Then, each participant will complete a self-reported questionnaire on their quality of life and level of physical activity. The remaining assessments of psychopathology, cognitive status and physical fitness will be guided and supervised by members of the research team.

- Stage 2: Longitudinal study of one prospective cohort with pre-post analysis. After this first phase, during the following 3 months, patients will be asked to complete a weekly record reflecting their mood, level of physical activity and medication changes (if applicable). A weekly reminder will be sent to each participant in the format chosen by each individual (message, e-mail or phone call) to complete the required information (through questionnaires in "Forms" format or verbally in the case of a phone call). During these weeks, they will be asked to take a one-week objective measurement of their daily physical activity. Those who accept will wear an accelerometer that will quantify their daily activity. Once the follow-up period is completed, the patients will be scheduled again for three new assessment sessions, in which the same tests and scales as in the previous phase will be executed.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years of age diagnosed with schizophrenia or schizoaffective disorder by a specialist physician.
2. be able to understand their involvement in the study when provided with the relevant information.
3. clinically stable, without behavioral disorganization that prevents participation in project activities and without suicidal ideation or suicide risk.
4. if they are under pharmacological treatment, they must be stable in the type of drug and its dosage and posology for at least 4 weeks.

Exclusion Criteria:

1. presenting pathologies that suppose a contraindication for the practice of supervised physical exercise (neurological diseases that suppose a cognitive deterioration such as to hinder the execution of tasks, musculoskeletal diseases that hinder stability and gait, or cardiovascular or metabolic diseases that suppose a risk for the individual).
2. being pregnant or in the puerperium period.
3. presenting in the last 3 months a moderate to severe comorbid substance abuse disorder that makes safe participation in the study impossible.
4. have been hospitalized for psychiatric or organic reasons in the 3 months prior to inclusion in the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of patients diagnosed with schizophrenia or schizoaffective disorder under follow-up in outpatient devices in the health area of Lugo.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The Modified Shuttle Walk Test (MSWT) | At baseline and after 3 months follow-up.
  requires the patient to walk/run a 10m course (delimited 0.5m from each end by a cone) at a speed that increases 0.6 km/h every minute. The start of the race is marked by a triple beep and each lap is indicated by a single beep. At the conclusion of each level, patients were instructed to increase their speed slightly and reminded that they were free to accelerate at any time during the test. The trial concluded under the following conditions: (1) the participant became too breathless to sustain the prescribed pace, (2) the participant deviated more than 0.5 m from the cone upon the beep, (3) the participant attained a heart rate exceeding 85% of their age-predicted maximum, or (4) in case the patient reported symptoms such as chest pain, angina, dizziness, mental confusion, or severe muscular exhaustion. With the meters performed in the test, we will estimate the maximum oxygen consumption (VO2max), using the formula proposed by Tous-Espelosin et al. in 2021.
The 5 repetitions Sit to Stand Test (5R STS) | At baseline and after 3 months follow-up.
  Participants will be instructed to sit in an armless chair of standard height (48 cm) with a hard seat, placed firmly against a wall. They will be required to cross their arms over their chest and keep their feet flat on the floor, wearing stable footwear throughout the test. Participants will be asked to stand up and sit down, landing firmly on the seat, five times as quickly as possible on the command "go". If the patient performs the test in 30 seconds or more, this time will be noted, and the test score will be recorded as 30 seconds. Using the Powerfrail app, the examiner will record the test performance on video to time the five repetitions, in addition to calculating the muscle power in W/kg.
The handgrip strength | At baseline and after 3 months follow-up.
  will be measured with a dynamometer (Takei model) following a standardized methodology developed by the University of Southampton in 2011, based on the recommendations of the American Society of Hand Therapists (ASHT). The patient will be seated in a chair with legs, backrest and arms fixed, forearms on the arms of the chair and wrist in neutral position with the thumb up. The patient will perform a measurement first with the right hand, then with the left hand and then repeat the procedure 2 more times. The best of the six measurements will be used for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Lucus Augusti, Lugo, Lugo, Spain